CLINICAL TRIAL: NCT05312840
Title: Efficacy and Safety of Conventional and Low-dose Platinum Gemcitabine Combined With Cindilimab With Delayed Administration in First-line Treatment of Advanced Squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: People's Hospital of Quzhou (Other)
Responsible Party: Principal Investigator, Jin Xuru, chief physician, People's Hospital of Quzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 320.6750.2021-02-135
Record Dates: First submitted 2022-03-14; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine dose group (Other): Routine dose group: Every three weeks as a cycle. On the first day of each cycle, Gemcitabine 1000mg / m2, Cisplatin 75mg / m2, Carboplatin auc5 were injected intravenously, and Gemcitabine 1000mg / m2 and Cindilimab 200mg were injected intravenously on the eighth day. After 4 or 6 cycles of treatment, if there is no disease progression, continue to use Cindilimab 200mg every three weeks until the disease progresses.
  Interventions: Drug: Cisplatin / Carboplatin，Gemcitabine，Cindilimab
- Low dose group (Other): Low dose group: Every three weeks as a cycle. Gemcitabine 750mg / m2, Cisplatin 56mg / m2 or Carboplatin auc3 were injected intravenously on the first day of each cycle 75. On the eighth day, Gemcitabine 750mg / m2 and Cindilimab 200mg were injected intravenously. After 4 or 6 cycles of treatment, if there is no disease progression, continue to use Cindilimab 200mg every three weeks until the disease progresses.
  Interventions: Drug: Cisplatin / Carboplatin，Gemcitabine，Cindilimab

INTERVENTIONS:
Drug: Cisplatin / Carboplatin，Gemcitabine，Cindilimab — 1. Routine dose group: Every three weeks as a cycle. On the first day of each cycle, Gemcitabine 1000mg / m2, Cisplatin 75mg / m2 / Carboplatin auc5 were injected intravenously, and Gemcitabine 1000mg / m2 and Cindilimab 200mg were injected intravenously on the eighth day; 2. Low dose group: every three weeks as a cycle. On the first day of each cycle, Gemcitabine 750mg / m2, Cisplatin 56mg / m2 / Carboplatin auc3 were injected intravenously 75. On the eighth day, Gemcitabine 750mg / m2 and Cindilimab 200mg were injected intravenously.

SUMMARY:
To observe the efficacy and safety of conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment of advanced squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
At present, Cindilimab combined with Gemcitabine and platinum chemotherapy has obtained the indication of first-line treatment for patients with advanced squamous non-small cell lung cancer, and has become one of the standard first-line treatment schemes for patients with advanced squamous non-small cell lung cancer. However, in DRIENT12 study, although it was confirmed that Cindilimab combined with Gemcitabine and platinum chemotherapy regimen can further delay or prevent the growth of cancer cells compared with placebo combined with Gemcitabine and platinum, in the process of treatment, due to serious adverse drug reactions, a considerable number of patients need to reduce the therapeutic dose of therapeutic drugs, and the body function of patients is damaged in this process, It will inevitably affect the treatment cycle, and even some patients stop treatment due to serious adverse drug reactions, and the serious adverse reactions of chemotherapy drugs will destroy the immune microenvironment, which will eventually affect the efficacy of the anti-cancer treatment. In addition, the mechanism of action of Cindilidone is different from that of chemotherapeutic drugs. It can kill tumor cells and inhibit tumor growth by activating human immune function. Therefore, in the combined scheme, reducing the dose of chemotherapy drugs to avoid too strong side effects damaging human immune function, destroying tumor cells to release antigens after the use of chemotherapy drugs, and continuing PD-1 monoclonal antibody to enhance human anti-tumor immunity may achieve the equivalent or better anti-tumor efficacy obtained in ORIENT12 research, and reduce treatment-related adverse reactions at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before implementing any test related process.
* Age ≥ 18 years old and ≤ 75 years old.
* Subjects with histologically or cytologically confirmed locally advanced (iiib-iiic), metastatic or recurrent (stage IV) squamous NSCLC (TNM lung cancer staging, 8th Edition, International Association for the study of lung cancer and Joint Committee on American Classification of cancer), inoperable and radical concurrent radiotherapy and chemotherapy, and who have not received systematic treatment before.
* The gene status is unknown, or the gene status of known histological specimens confirms that there is no EGFR gene sensitive mutation or ALK gene fusion mutation.
* According to the evaluation criteria of solid tumor efficacy (RECIST v1.1), at least one lesion can be measured by imaging. Lesions located in the radiation field of previous radiotherapy can be regarded as measurable lesions if they are confirmed to have progression.
* Have not received any systematic antitumor treatment for advanced / metastatic diseases in the past. Subjects who have previously received platinum containing adjuvant / neoadjuvant chemotherapy or radical chemoradiotherapy for advanced diseases, if the interval between disease progression or recurrence and the end of the last chemotherapeutic drug treatment is at least 6 months, are allowed to be included in this study.
* Subjects with brain metastases who are asymptomatic or have stable symptoms after local treatment are allowed to be included as long as they meet the following conditions: 1) measurable lesions outside the central nervous system, 2) no symptoms of the central nervous system or no aggravation of symptoms for at least 2 weeks, 3) no glucocorticoid treatment is required, or glucocorticoid treatment is stopped within 7 days before the first administration, Or the dosage of glucocorticoid is stable and reduced to less than 10mg / day prednisone (or equivalent dose) within 7 days before the first administration.
* Patients were allowed to receive palliative radiotherapy, but the end time of radiotherapy was 7 days before the administration of the first study drug, and the toxicity related to radiotherapy recovered to less than or equal to grade 1 (CTCAE V5.0).
* ECoG score: 0-1.
* Expected survival time > 3 months.
* For adequate organ function, the subjects shall meet the following laboratory indexes: 1) the absolute value of neutrophils (ANC) ≥ 1.5x109/l without granulocyte colony stimulating factor in recent 14 days; 2) Platelets ≥ 100 without blood transfusion in recent 14 days × 109/L 3) Hemoglobin > 9g / dl without blood transfusion or erythropoietin in recent 14 days; 4) Total bilirubin ≤ 1.5 times the upper limit of normal value (ULN) 5) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤ 2.5 times ULN (ALT or AST ≤ 5 is allowed for subjects with liver metastasis × ULN） 6) Serum creatinine ≤ 1.5 times ULN and creatinine clearance rate (calculated by Cockcroft Gault formula) ≥ 60 ml / min; 7) Good coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; 8) Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is beyond the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled; 9) The myocardial enzyme spectrum is within the normal range (for example, simple laboratory abnormalities that are not clinically significant according to the comprehensive judgment of the researcher are also allowed to be included in the group).
* For female subjects of childbearing age, urine or serum pregnancy test shall be conducted within 3 days before receiving the first study drug administration (day 1 of cycle 1) and the result is negative. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non childbearing age are defined as having been postmenopausal for at least 1 year or having undergone surgical sterilization or hysterectomy.
* If there is a risk of pregnancy, all subjects (male or female) are required to use contraceptives with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last study drug administration (or 180 days after the last study drug administration).

Exclusion Criteria:

* Pathology is adenocarcinoma or small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC.
* Received radiotherapy before administration of the first study drug, Meet one of the following conditions: 1) more than 30% of bone marrow had received radiotherapy within 14 days before treatment; 2) received radiotherapy for lung lesions within 6 weeks before treatment and the dose was > 30Gy (the enrolled subjects must recover from the toxicity of previous radiotherapy to grade 1 or below, do not need glucocorticoid treatment and have no history of radiation pneumonia) 3) The end time of palliative radiotherapy was within 7 days before the administration of the first study drug.
* Other malignant diseases other than NSCLC diagnosed within 5 years before the first administration (excluding radical skin basal cell carcinoma, skin squamous epithelial carcinoma, and / or radical resection of carcinoma in situ).
* Currently participating in intervention clinical research treatment, or receiving other research drugs or using research instruments within 4 weeks before the first administration.
* Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or co inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137).
* Received systemic treatment with Chinese patent medicine with anti NSCLC indications or drugs with immunomodulatory effect (including thymosin, interferon and interleukin, except for local use to control pleural effusion) within 2 weeks before the first administration.
* Active autoimmune diseases requiring systemic treatment (such as the use of disease relief drugs, glucocorticoids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (such as thyroxine, insulin or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatment.
* Being treated with systemic glucocorticoids (excluding nasal spray, inhaled or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first administration of the study; Note: it is allowed to use glucocorticoids in physiological doses (≤ 10 mg / day prednisone or equivalent).
* There is clinically uncontrollable pleural effusion / peritoneal effusion (subjects who do not need to drain effusion or stop drainage for 3 days and have no significant increase in effusion can be enrolled).
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
* Those who are known to be allergic to active ingredients or excipients such as cindilimab, pemetrexed, gemcitabine, carboplatin and cisplatin.
* Not fully recovered from toxicity and / or complications caused by any intervention before starting treatment (i.e. ≤ grade 1 or reaching baseline, excluding fatigue or hair loss).
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1 / 2 antibody positive).
* untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number at the same time was higher than the upper limit of normal value in the laboratory of the research center). Note: hepatitis B patients who met the following criteria can also be admitted into the group: 1) HBV viral load <1000 copy /ml (200 IU/ml) before the first dose, the subjects should receive anti HBV therapy to avoid reactivation of the virus during the whole course of chemotherapy (2). Subjects with anti HBc (+), HBsAg (-), anti HBs (-) and HBV viral load (-), Prophylactic anti HBV treatment is not required, but virus reactivation needs to be closely monitored.
* Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the lower limit of detection).
* Have received live vaccine within 30 days before the first administration (cycle 1, day 1); Note: it is allowed to receive inactivated virus vaccine for injection against seasonal influenza within 30 days before the first administration; However, live attenuated influenza vaccines administered intranasal are not allowed.
* Pregnant or lactating women.
* There are any serious or uncontrollable systemic diseases, such as: 1) there are significant abnormalities in rhythm, conduction or morphology of resting ECG and the symptoms are serious and difficult to control, such as complete left bundle branch block, heart block above grade II, ventricular arrhythmia or atrial fibrillation; 2) Unstable angina pectoris, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) grade ≥ 2; 3) Myocardial infarction occurred within 6 months before enrollment; 4) Poor blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); 5) A history of noninfectious pneumonia requiring glucocorticoid treatment within 1 year before the first administration, or the current presence of clinically active interstitial lung disease; 6) Active pulmonary tuberculosis; 7) There are active or uncontrolled infections requiring systemic treatment; 8) There were clinically active diverticulitis, abdominal abscess and gastrointestinal obstruction; 9) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; 10) poor control of diabetes (fasting blood glucose (FBG) > 10mmol/L). 11) Urine routine examination showed that urinary protein was ≥ + +, and the 24-hour urinary protein was confirmed to be more than 1.0 g; 12) Subjects with mental disorders and unable to cooperate with treatment.
* There is no evidence that the participants in the study group have abnormal medical history or other potential conditions that may hinder the study group from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The objective response rate (ORR) of treatment was evaluated according to RECIST (v1.1). | 36 months
  To evaluate the objective response rate (ORR) of subjects with advanced squamous non-small cell lung cancer treated with conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment. ORR is defined as the proportion of subjects with complete response (CR) and partial response (PR) in the total subjects.
Assess the subject's progression free survival (PFS) according to RECIST (v1.1). | 36 months
  To evaluate the progression free survival (PFS) of subjects with advanced squamous non-small cell lung cancer treated with conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment. PFS is defined as the time from the beginning of treatment to the first imaging disease progression or death, whichever occurs first.
Assess the subject's disease control rate (DCR) according to RECIST (v1.1). | 36 months
  To evaluate the disease control rate (DCR) of subjects with advanced squamous non-small cell lung cancer treated with conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment. DCR is defined as the proportion of total subjects with complete remission (CR), partial remission (PR) and disease stability (SD).
The duration of remission (DOR) was assessed according to RECIST (v1.1). | 36 months
  To evaluate the duration of remission (DOR) of subjects with advanced squamous non-small cell lung cancer treated with conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment. DOR is defined as the time interval from the first recorded remission to disease progression or death, whichever occurs first.
The overall survival (OS) of the subjects was evaluated according to RECIST (v1.1). | 36 months
  To evaluate the overall survival (OS) of subjects with advanced squamous non-small cell lung cancer treated with conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment. OS is defined as the time from the beginning of treatment to the death of subjects from any cause.

SECONDARY OUTCOMES:
The incidence of adverse events was evaluated according to NCI CTCAE (v5.0). | 36 months
  To evaluate the incidence of adverse events in subjects with advanced squamous non-small cell lung cancer treated with conventional and low-dose platinum Gemcitabine combined with Cindilimab with delayed administration in first-line treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xuru Jin, Principal Investigator — People's Hospital of Quzhou
Locations (1):
- Quzhou people's Hospital, Quzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No